CLINICAL TRIAL: NCT04497220
Title: Will Negative Phrasing Create a Nocebo Effect During Epidural Placement When Compared to Positive Phrasing? A Randomized Controlled Trial
Brief Title: Poke and a Placebo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANES-2020-29006
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia
Keywords: Epidural Anesthesia (labor)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nocebo Group (Placebo Comparator): Participants in this group will receive the control treatment
  Interventions: Behavioral: Negative Connotation Langauge
- Positive Connotation Group (Experimental): Participants in this group will receive the experimental treatment.
  Interventions: Behavioral: Positive Connotation Language

INTERVENTIONS:
Behavioral: Negative Connotation Langauge — The study intervention consists of two separate scripts read to the patient by the anesthesiologist performing their labor epidural. The control script includes language containing the wording "Poke and a burn" said prior to numbing medication for the epidural procedure. There will be no difference in the epidural placement, medications, or the rest of the script.
  Arms: Nocebo Group
Behavioral: Positive Connotation Language — The study intervention consists of two separate scripts read to the patient by the anesthesiologist performing their labor epidural. The experimental script includes language containing the wording "this is numbing medication, which will make the rest of the procedure go easier" said prior to numbing medication for the epidural procedure. There will be no difference in the epidural placement, medications, or the rest of the script.
  Arms: Positive Connotation Group

SUMMARY:
To discover if a positive description of the procedure for an epidural can reduce the overall pain score associated with the procedure.

DETAILED DESCRIPTION:
The study intervention consists of two separate scripts read to the patient by the anesthesiologist performing their labor epidural. One script will contain the wording "Poke and a burn" prior to subcutaneous local anesthetic administration for the epidural placement and one will contain "this is numbing medication, which will make the rest of the procedure go easier". There will be no difference in the epidural placement, medications, or the rest of the script.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy
* requesting an epidural for the first time

Exclusion Criteria:

* previous epidural (either for labor or for surgery)
* BMI greater than 40 kg/m^2
* previous lumbar spine surgery
* inability to speak English
* a history of chronic pain or are on chronic opioids
* a history of opioid drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Max pain score during the epidural procedure | 1 hour
  Maximum pain score will be measured using a single 11-point Numeric Rating Scale 0-10, where 0 is no pain and 10 is maximum imaginable pain.

SECONDARY OUTCOMES:
Overall satisfaction during the epidural procedure | 1 hour
  Overall satisfaction during the epidural procedure will be measured used a 5-point likert scale: 5=very satisfied, 4=satisfied, 3=neither satisfied or dissatisfied, 2=dissatisfied, 1=very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Berg, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States